CLINICAL TRIAL: NCT05575115
Title: Non-Inferiority of Peer Comparison Interventions vs. Control Condition in BEARI Trial
Brief Title: Non-Inferiority of Peer Comparison Interventions
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Other Study IDs: HS-11-00249; 1RC4AG039115 (NIH)
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Tract Infections
Keywords: Antibiotics; Inappropriate Prescribing; Behavioral Research
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peer Comparison: Providers from the BEARI trial who received the Peer Comparison intervention.
  Interventions: Behavioral: Peer Comparison
- Control: Providers from the BEARI trial who did not receive the Peer Comparison intervention.

INTERVENTIONS:
Behavioral: Peer Comparison — Peer comparison was an email-based intervention. Clinicians were ranked from highest to lowest inappropriate prescribing rate within each region using EHR data. Clinicians with the lowest inappropriate prescribing rates (the top-performing decile) were told via monthly email they were "Top Performers". The remaining clinicians were told that they were "Not a Top Performer" in an email that included the number and proportion of antibiotic prescriptions they wrote for antibiotic-inappropriate acute respiratory tract infections, compared with the proportion written by top performers.
  Groups: Peer Comparison

SUMMARY:
The objective of this study is to test the hypothesis that the Peer Comparison intervention in the Use of Behavioral Economics to Improve Treatment of Acute Respiratory Infections (BEARI) trial (Meeker et al. 2016) promoting antibiotic stewardship did not adversely impact physician job satisfaction as measured in the study exit survey at trial completion. Detrimental impacts on job satisfaction is a phenomenon that was observed in a randomized controlled trial using a Peer Comparison intervention with different characteristics from the BEARI trial. (Reiff et al. 2022) The BEARI trial sample size, intraclass correlation, and measurement of job satisfaction are comparable to Reiff et al. 2022.

DETAILED DESCRIPTION:
This secondary analysis includes all providers from the Use of Behavioral Economics to Improve Treatment of Acute Respiratory Infections (BEARI) trial who completed the exit survey following 18 month trial completion. The objective of this study is to test the hypothesis that the Peer Comparison intervention in the BEARI trial (Meeker et al. 2016) promoting antibiotic stewardship did not adversely impact physician job satisfaction. Detrimental impacts on job satisfaction is a phenomenon that was observed in a randomized controlled trial using a Peer Comparison intervention with different characteristics from the BEARI trial. (Reiff et al. 2022) The BEARI trial sample size, intraclass correlation, and measurement of job satisfaction are comparable to Reiff et al. 2022.

The differences in Peer Comparison interventions between BEARI and Reiff et al. include the following:

1. Differences in physicians' control and agency over patient adherence to screening recommendations vs. their own antibiotic prescribing
2. Relatedly, in the antibiotic stewardship study, there were achievable benchmarks for improvement, including a feedback and ranking framework allowing all physicians to attain the highest status and thus obtain positive feedback.
3. Differences in framing and presentation of messages

The investigators define a clinically significant detrimental effect on job satisfaction as 27% of individuals reducing job satisfaction ratings by one point on a 5-point likert scale. This shift is equivalent to a mean difference of 0.32 and a Cohen's d of 0.36. This difference corresponds to approximately a ⅓ reduction in job satisfaction on a 5-point likert scale.

H0: The BEARI Peer Comparison intervention had a clinically and statistically significant detrimental effect on physician job satisfaction. Control-PeerComparison>=0.32

HA: The Peer Comparison intervention had no clinically significant negative impact on physician job satisfaction. Control-PeerComparison<0.32

The investigators will conduct a traditional hypothesis test Control-PeerComparison= 0.0 as a secondary analysis.

ELIGIBILITY:
Inclusion Criteria:

* All providers included in the BEARI trial

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all providers in the BEARI trial. The intent of the BEARI trial was to apply behavioral economic theory to reduce the rate of antibiotic prescriptions for acute respiratory diagnoses for which guidelines do not call for antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Job satisfaction | 18 months
  Impact of BEARI Peer Comparison intervention on Job Satisfaction, as measured by the following question completed as part of the BEARI trial exit survey: "Please indicate how much you agree or disagree with the following statement. Overall, I am satisfied with my current job."

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California

REFERENCES:
- [Background] Persell SD, Friedberg MW, Meeker D, Linder JA, Fox CR, Goldstein NJ, Shah PD, Knight TK, Doctor JN. Use of behavioral economics and social psychology to improve treatment of acute respiratory infections (BEARI): rationale and design of a cluster randomized controlled trial [1RC4AG039115-01]--study protocol and baseline practice and provider characteristics. BMC Infect Dis. 2013 Jun 27;13:290. doi: 10.1186/1471-2334-13-290. PMID 23806017
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Background] Reiff JS, Zhang JC, Gallus J, Dai H, Pedley NM, Vangala S, Leuchter RK, Goshgarian G, Fox CR, Han M, Croymans DM. When peer comparison information harms physician well-being. Proc Natl Acad Sci U S A. 2022 Jul 19;119(29):e2121730119. doi: 10.1073/pnas.2121730119. Epub 2022 Jul 14. PMID 35858307
- [Derived] Doctor JN, Goldstein NJ, Fox CR, Linder JA, Persell SD, Stewart EP, Knight TK, Meeker D. Clinician Job Satisfaction After Peer Comparison Feedback: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317379. doi: 10.1001/jamanetworkopen.2023.17379. PMID 37289454